CLINICAL TRIAL: NCT00119834
Title: Interagency Registry for Mechanically Assisted Circulatory Support (Intermacs)
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1296; N01-HV-18246 (Other: NHLBI)
Record Dates: First submitted 2005-07-06; First posted 2005-07-14 (Estimated); Last update posted 2018-04-09 (Actual); Status verified 2018-04

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Heart Failure, Congestive
Keywords: Heart Failure; Intermacs; Pedimacs; Mechanical Circulatory Support; Ventricular Assist Device
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Biospecimen Retention: Samples With DNA — DNA sample collection was an optional portion of the project during the first contract period (2005-2010). Tissue and Blood specimens were collected at the time of implant, explant or exchange of the mechanical circulatory assist device. Intermacs no longer collects blood or tissue specimens.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Mechanical Circulatory Support Device (MCSD) — INTERMACS is an observational registry of adult and pediatric patients with end stage heart failure that receive a legally utilized Mechanical Circulatory Support Device.

SUMMARY:
The Intermacs registry is a national quality improvement system designed to advance the understanding and application of mechanical circulatory support in order to improve the duration and quality of life in patients with advanced heart failure.

DETAILED DESCRIPTION:
Background:

Over the last several decades, MCSDs have been developed to augment or supplant failing myocardial performance. This therapy has been used successfully as a bridge to heart transplantation, a bridge to recovery, and as permanent implantation or "destination therapy" for intractable heart failure. Although heart transplantation offers life-saving therapy for selected patients, its use is limited by a supply of donor organs that currently meets less than one-tenth the need. As a consequence, the number of MCSD implantations has increased in recent years.

Despite favorable survival and quality of life outcomes, MCSDs do have severe and sometimes life-threatening complications, including infection, thrombosis, and device failure. The development of new procedures and devices to reduce these complications will be expedited by the work of the registry involving the systematic, independent analysis of MCSD implantation procedures and outcomes. The National Heart, Lung, and Blood Institute (NHLBI) will collaborate with the Centers for Medicare and Medicaid Services (CMS) and the Food and Drug Administration (FDA) in monitoring the work of the registry to permit the development of standard reporting of patient characteristics, indications, implantation procedures, and adverse events.

Intermacs Design Narrative:

The goals of the registry include the following:

1. Develop standard methods to collect data used to characterize heart failure patients receiving MCSDs, and develop methods of collecting demographic data of device use patient outcomes
2. Collect, process, and store patients' clinical data
3. Analyze collected data
4. Provide these resources to researchers outside the registry
5. Publish and disseminate results

Intermacs has included pediatric patients since the inception of the registry in 2006 with an increased effort in September 2012 to include pediatric subjects. This focus is called Pedimacs. Pedimacs utilizes the Intermacs protocol. Due to collection of pediatric-only data elements, a separate Users' Guide has been developed for Pedimacs.

Intermacs now serves as the national quality improvement system to assess the characteristics, treatments and outcomes of patients receiving legally utilized mechanical circulatory support devices. The protocol has undergone several changes since its inception in 2006. The Current protocol (Protocol 5.0) reflects the latest changes and the necessity for a waiver of informed consent and authorization for participants.

In January 2013 the Medical Arm of the Interagency Registry for Mechanically Assisted Circulatory Support (Medamacs) was established to capture data on patients with advanced heart failure who were not receiving mechanical circulatory support devices. The aims of Medamacs are to:

1. Identify prospectively a population of ambulatory patients on optimal medical therapy for whom chronic heart failure limits both function and survival to a range where elective implantation of left ventricular assist devices should offer meaningful benefit.
2. Design an integrated endpoint of survival and objective functional assessment that provides more discrimination between chronic ambulatory heart failure and current device outcomes than survival alone.
3. Evaluate patient perceptions about their cardiac condition, ventricular assist device technology, preferences for their care, and thresholds for considering device implant.

Enrollment in Medamacs has closed.

The clinicaltrials.gov identification number for Medamacs is NCT01932294.

ELIGIBILITY:
Inclusion Criteria:

* Legally utilized MCSD implanted on or after March 1, 2006; every consented patient who receives an eligible MCSD at a participating center will be enrolled, regardless of reason (i.e., bridge-to-recovery, bridge-to-alternative bridge, bridge-to-clinical improvement for transplant eligibility, bridge-to-transplant, destination therapy). Beginning June 1, 2014, and with lnstitutional Review Board approval, participating sites may enroll patients under a waiver of informed consent and authorization.
* Eligible devices include all of the following: 1) approved devices for any indications; 2) Intermacs-linked trial of investigational device or approved device for investigational indications, for which data will be entered via the Intermacs framework; 3) external trial of investigational device or approved device for investigational indications, for which data will be collected by an external group; 4) compassionate use of investigational devices or approved devices outside of approved indications or clinical trials

Exclusion Criteria:

* Currently incarcerated

Min Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with end-stage heart failure that receive a legally utilized mechanical circulatory support device.
Sampling Method: Non-Probability Sample
Enrollment: 23472 (Actual)
Dates: Start 2005-06 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Collect and analyze clinical and laboratory data from patients who are receiving mechanical circulatory support devices (MCSD) for end-stage heart failure. | Collected as part of the registry

CONTACTS AND LOCATIONS:
Overall Officials: James K. Kirklin, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) is not available. De-identified datasets may be available upon approval.

REFERENCES:
- [Derived] Brisco MA, Kimmel SE, Coca SG, Putt ME, Jessup M, Tang WW, Parikh CR, Testani JM. Prevalence and prognostic importance of changes in renal function after mechanical circulatory support. Circ Heart Fail. 2014 Jan;7(1):68-75. doi: 10.1161/CIRCHEARTFAILURE.113.000507. Epub 2013 Nov 8. PMID 24214901